CLINICAL TRIAL: NCT02243566
Title: Morning Hypertension and Patient Self-monitoring
Brief Title: Post-marketing Surveillance Study With MicardisPlus® in Treatment of Morning Hypertension (Self-monitored by Patient)
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 502.513
Record Dates: First submitted 2014-09-16; First posted 2014-09-18 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — telmisartan, hydrochlorothiazide drug combination; Telmisartan; Hydrochlorothiazide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Essential hypertension
  Interventions: Drug: MicardisPlus®

INTERVENTIONS:
Drug: MicardisPlus®
  Other Names: Telmisartan in combination with hydrochlorothiazide

SUMMARY:
The purpose of the study was to examine the effect of six- to eight-week treatment with MicardisPlus® on blood pressure and the effect of patient self-monitoring on blood pressure control. In addition, the post-marketing surveillance study offered the possibility to obtain information about the influence on different laboratory parameters during treatment with MicardisPlus® from an unselected patient group under office conditions

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Hypertension

Exclusion Criteria:

* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients with essential hypertension
Sampling Method: Non-Probability Sample
Enrollment: 2707 (Actual)
Dates: Start 2006-04; Primary Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Changes in morning blood pressure (systolic and diastolic) | Pre-dose, up to 8 weeks after start of treatment
Changes from baseline in laboratory values | Pre-dose, up to 8 weeks after start of treatment
Investigator assessment of efficacy on a 5-point scale | Up to 8 weeks after start of treatment
Investigator assessment of influence on metabolism on a 3-point scale | Up to 8 weeks after start of treatment
Investigator assessment of tolerability on a 5-point scale | Up to 8 weeks after start of treatment
Number of patients with adverse events | Up to 8 weeks